CLINICAL TRIAL: NCT01637103
Title: Treatment of Depressive Symptoms in Breast Cancer Patients: Comparison of Cognitive Therapy and Bright Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Josée Savard, Professeure titulaire/Chercheuse, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H10-12-123
Record Dates: First submitted 2012-04-18; First posted 2012-07-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Treatment of Depressive Symptoms in Cancer Patients
Keywords: Cancer; Depression; Anxiety; Fatigue; Sleep; Quality of life; Cognitive therapy; Bright light therapy
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders; Fatigue | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive therapy of depression (Experimental)
  Interventions: Behavioral: Cognitive therapy of depression
- Bright light therapy (Experimental)
  Interventions: Behavioral: Bright light therapy
- Waiting list (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive therapy of depression — Cognitive therapy will involve eight individual weekly sessions of 50 minutes with a Ph.D. student in psychology.
  Arms: Cognitive therapy of depression
Behavioral: Bright light therapy — Bright light therapy will consist of a 30-min daily morning exposition to a 10 000-lux BLT lamp during 8 weeks.
  Arms: Bright light therapy

SUMMARY:
Depressive symptoms are highly frequent among cancer patients. These symptoms significantly impair quality of life (e.g., hopelessness, greater risk of suicidal behaviours) and may even affect patients' prognosis (e.g., through decreased adherence to cancer treatments). Cognitive therapy (CT) is an established treatment for depression in the general population, but its efficacy has not yet been investigated in non-metastatic cancer patients. Furthermore, because the accessibility to CT is very limited in routine cancer care and because many patients are reluctant to use pharmacological treatment, they often turn to alternative treatments such as bright light therapy (BLT), but empirical data on its efficacy are needed before its use can be recommended. Goal 1: To assess at post-treatment, as compared to a waiting-list control condition, the effect of bright light therapy (BLT) and cognitive therapy (CT): (1a) in reducing depressive symptoms; and (1b) in improving subjective and objective sleep parameters, in reducing fatigue and anxiety and in increasing patients' functioning and quality of life. Goal 2: To compare at post-treatment and at 3- and 6-month follow-ups the effect of BLT and CT : (2a) in reducing depressive symptoms; and (2b) in improving subjective and objective parameters of sleep, in reducing fatigue and anxiety and in increasing patients' functioning and quality of life. It is hypothesized that, As compared to control patients after their waiting period, both BLT and CT groups will have significantly greater improvement of all symptoms at post-treatment. However, as compared to BLT patients, CT patients will show greater improvements of all symptoms at post-treatment and at 3- and 6-month follow-ups. This study will provide empirical data on the efficacy of two approaches for treating depressive symptoms in cancer patients in order to better inform the scientific community, health care providers, and patients on the most effective depression treatments to implement in cancer care.

ELIGIBILITY:
Inclusion Criteria:

* having received a diagnosis for a stage I-III cancer within the past 18 months;
* having a score of 7 or higher on the depression subscale of the Hospital Anxiety and Depression Scale (HADS-D)84 or of 14 or higher on the Beck Depression Inventory-II (BDI-II);

Exclusion Criteria:

* have received bright light therapy in the past month or having previously received cognitive therapy for depression;
* having severe cognitive impairments (e.g., diagnosis of Parkinson's disease, dementia, or Mini-Mental State Examination [MMSE] score < 27);
* meeting DSM-IV criteria for a major depressive episode of severe intensity, or another severe psychiatric disorder (e.g., psychotic, bipolar, or substance use disorder);
* presenting suicidal ideations with a risk of acting out, or having attempted suicide in the past five years;
* having started a new psychotropic medication or having modified the dosage or frequency of use during the past two weeks;
* currently taking a photosensitive medication (e.g., lithium, L-tryptophan);
* having evidence of an ocular pathology from an optometrist exam or a medical condition contraindicating the use of bright light therapy (e.g., severe cataracts, glaucoma, diabetes).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms | Pre-treatment (at recruitment; about 2 weeks before starting the experimental condition of 8 weeks), post-treatment (immediately after the experimental condition of 8 weeks), 3-month follow-up and 6-month follow-up

SECONDARY OUTCOMES:
Changes in subjective and objective parameters of sleep | Pre-treatment (at recruitment; about 2 weeks before starting the experimental condition of 8 weeks), post-treatment (immediately after the experimental condition of 8 weeks), 3-month follow-up and 6-month follow-up
Changes in fatigue | Pre-treatment (at recruitment; about 2 weeks before starting the experimental condition of 8 weeks), post-treatment (immediately after the experimental condition of 8 weeks), 3-month follow-up and 6-month follow-up
Changes in anxiety | Pre-treatment (at recruitment; about 2 weeks before starting the experimental condition of 8 weeks), post-treatment (immediately after the experimental condition of 8 weeks), 3-month follow-up and 6-month follow-up
Changes in quality of life | Pre-treatment (at recruitment; about 2 weeks before starting the experimental condition of 8 weeks), post-treatment (immediately after the experimental condition of 8 weeks), 3-month follow-up and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Josée Savard, Ph.D., Study Director — Laval University Cancer Research Center
Locations (1):
- L'Hôtel-Dieu de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Desautels C, Savard J, Ivers H. Moderators of Cognitive Therapy and Bright Light Therapy Effects on Depressive Symptoms in Patients with Breast Cancer. Int J Behav Med. 2019 Aug;26(4):380-390. doi: 10.1007/s12529-019-09802-6. PMID 31264101
- [Derived] Desautels C, Savard J, Ivers H, Savard MH, Caplette-Gingras A. Treatment of depressive symptoms in patients with breast cancer: A randomized controlled trial comparing cognitive therapy and bright light therapy. Health Psychol. 2018 Jan;37(1):1-13. doi: 10.1037/hea0000539. Epub 2017 Nov 27. PMID 29172605